CLINICAL TRIAL: NCT06698601
Title: Impact of Wild Blueberries (Vaccinium Myrtillus) on the Intestinal Barrier, Microbiome and Inflammation in Chronic Colitis - a Prospective Randomized Crossover Study
Brief Title: Wild Blueberries in Colitis
Acronym: BlueVantage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: UniversitÃ¤t Duisburg-Essen (Unknown); German Crohn's and Colitis Association (DCCV e.V.) (Unknown); Wilhelm Doerenkamp Foundation (Unknown)
Responsible Party: Principal Investigator, Jost Langhorst, Univ. Prof. Dr. med, Universität Duisburg-Essen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23068
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis (UC); Crohn Disease (CD)
Keywords: ulcerative colitis; crohn disease; integrative medicine; intestinal barrier; inflammatory bowel disease; confocal laser endomicroscopy; wild blueberry; bilberry; nutrition; microbiome; inflammation; chronic colitis
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: All participants undergo both study arms. This means that each participant is in the blueberry (intervention) group for a period of 3 months and is in the control group for 3 months. The order in which the participants receive the forms of therapy is determined randomly. Thus, half of the study participants start the supplementary blueberry intake directly after the inpatient stay, the second half three months later (crossover design).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): wild blueberry
  Interventions: Dietary Supplement: blueberry-rich diet
- Control group (Other): No wild blueberry
  Interventions: Other: Control diet

INTERVENTIONS:
Dietary Supplement: blueberry-rich diet — The study participants follow a diet rich in blueberries for 12 weeks based on the nutritional therapy and the integrative medical concept taught during their inpatient stay at the clinic for internal and integrative medicine in Bamberg.
  Participants will drink approximately 35g of a powder made from wild, freeze-dried blueberries containing 780mg of anthocyanines stirred in a glas of water every morning for a period of 12 weeks.
  Arms: Intervention group
Other: Control diet — The study participants will focus on the nutritional therapy and the integrative medical concept taught during their inpatient stay at the clinic for internal and integrative medicine in Bamberg.
  Participants will receive no additional blueberry treatment.
  Arms: Control group

SUMMARY:
The goal of this exploratory, prospective, monocentric randomized crossover study is to investigate the influence of a blueberry-rich diet compared to a blueberry-poor diet on the microbiome, the intestinal barrier and the inflammatory process in IBD patients with chronic colitis.

The main question the study aims to answer is:

* Does a diet rich in blueberries compared to a diet low in blueberries have an influence on disease activity, intestinal inflammation and symptoms in IBD patients with chronic colitis?

Ulcerative Colitis (UC) and Crohn's disease (MC) patients are recruited during an inpatient stay at the Clinic for Internal and Integrative Medicine in Bamberg, Germany. During their routine inpatient stay, patients are treated by an interdisciplinary team using a comprehensive multimodal integrative inpatient therapy concept that combines conventional medicine with a wide range of integrative non-pharmacological treatments, phytotherapy, lifestyle-modification and nutritional therapy. During this time, it is verified whether the patients can participate in the study.

The study consists of two study arms, which are conducted in a cross-over design:

* Intervention arm: in this study arm, participants receive 12 weeks of blueberry therapy in addition to the regular two weeks of inpatient care at the Clinic for Internal and Integrative Medicine in Bamberg. The blueberry therapy includes drinking around 35 g of blueberry powder stirred into water once a day for 12 weeks.
* Control arm: in this study arm, participants receive the standard therapy (integrative medical therapy concept described above) during the regular two-week hospital stay. There is no additional blueberry intake.

Due to the crossover study design, all participants undergo both study arms. This means that each participant takes the supplementary blueberry powder (intervention) for a period of 3 months and the control therapy for 3 months. The order in which the participants receive the forms of therapy is determined randomly. Thus, half of the study participants start the supplementary blueberry intake directly after the inpatient stay, the second half three months later (cross-over principle).

UC and MC patients will:

* initially receive a clinically indicated colonoscopy with confocal laser endomicroscopy (CLE) during their routine inpatient stay at the Clinic for Internal and Integrative Medicine in Bamberg
* return to the clinic for an optional sigmoidoscopy with CLE after 12 and 24 weeks
* answer questionnaires at study start as well as after 12 and 24 weeks to analyze their quality of life, the severity of their symptoms and their disease activity
* give samples of blood, urine, stool and bile fluid as well as intestinal biopsies during the colonoscopy/sigmoidoscopy at study start as well as after 12 and 24 weeks
* document their intake of blueberry powder as well as their symptoms and stool frequencies in a diary throughout the study participation

DETAILED DESCRIPTION:
Background:

Chronic inflammatory bowel disease (IBD) affects the lives of millions of people worldwide due to recurrent, severe clinical symptoms, potential complications and ongoing medical interventions. The scientific community currently assumes a multicausal pathogenesis in IBD caused by an unfavorable constellation of genetic predisposition, imbalance of pathogenic to symbiotic gut bacteria (dysbiosis) and harmful environmental and lifestyle factors resulting in an excessive immune response.

The intestinal barrier and the microbiome play a key role in maintaining intestinal balance and health. The intestinal barrier protects our body from bacteria, viruses and fungi in the intestinal lumen, while it enables the absorption of nutrients at the same time. In case of a leaky gut, microbial pathogens or their components can enter the deeper cell layers of the intestine and cause acute and long-term inflammatory reactions. The composition of the gut microbiome, i.e. the community of billions of microorganisms living in the gut, has a significant influence on the intestinal barrier and gut health. Beneficial bacteria stabilize the intestinal barrier, strengthen local defenses (mucin and IgA production) and inhibit pro-inflammatory immune reactions and cell death. In contrast, harmful bacteria (pathobionts) disrupt the intestinal barrier, dysregulate cell death and proliferation, which leads to the release of pro-inflammatory signaling substancesand and an immune response causing inflammation.

While previous attempts to develop pharmacological therapies to improve gut barrier function have been unsuccessful, an increasing number of preclinical and clinical trial results highlight the significant impact of a plant-based diet through its modulatory effect on the gut microbiome and the gut barrier in IBD. However, further research is needed to evaluate the role of individual dietary components and complex dietary interventions with anti-inflammatory potential in the prevention and treatment of IBD.

The high levels of prebiotic food components in a plant-rich diet are of particular importance in the treatment of intestinal barrier disorders and the microbiome.

Preclinical and clinical studies highlight the modulatory effect of berries, especially blueberries (Vaccinium myrtillus), on the microbiome, gut health and inflammation due to their richness in prebiotically active polyphenols, flavonoids, anthocyanins and fiber.

However, the influence of blueberries on the intestinal barrier and the microbiome in colitis patients has not yet been investigated. Mechanistically oriented clinical studies are needed to confirm the prebiotic and preclinical findings in the clinic. Through a targeted combination of clinical testing on patients, ex vivo examination of biopsy material and cell biological studies at protein and transcriptome level, it should be possible to develop a comprehensive picture of the influence of a blueberry-rich diet, but also of the underlying pathomechanisms affected.

Aim of the study:

Determination of the influence of a three-month blueberry-rich diet compared to a diet with a low blueberry content on disease activity, intestinal inflammation and symptoms in patients with chronic colitis - initiated as part of a routine inpatient stay during which patients are treated with a comprehensive multimodal integrative therapy concept with dietary changes.

Exploratory study design:

This is an exploratory, prospective, monocentric, randomized, crossover study. 60 IBD patients are randomized into two groups of 30 subjects each. During a period of 6 months, which follows the inpatient-initiated integrative medical lifestyle modification program, participants undergo two consecutive phases of 3 months each marked by a blueberry-rich and a blueberry-poor diet. Dependent on the study group, half of the study participants start the supplementary blueberry intake directly after the inpatient stay, the second half three months later (cross-over principle).

Before the start of the study (W0), the colon of the participants is initially examined for macroscopic inflammation and for intestinal barrier disorders using confocal laser endomicroscopy as part of regular inpatient care. In order to investigate the influence of the integrative therapy with or without blueberry intake on the intestinal barrier and colonic inflammation, this will be checked after the end of the first 3 months (W12) and after 6 months (W24) in a voluntary control sigmoidoscopy with confocal laser endomicroscopy (CLE) as part of a short inpatient stay.

During the endoscopy, biopsies, bile, stool, urine and blood samples important for the study are taken for examination. These serve to clarify mechanistic relationships between the intestinal barrier function, the microbiome, its metabolic products (metabolome), the immune system, the oxidative stress profile, the antioxidative capacity and the inflammatory process (inflammation markers, immune cells and cytokines). In addition, participants will receive questionnaires at all three time points (W0, W12, W24) to evaluate their IBD-specific and general quality of life, symptoms, disease activity, fatigue and stress levels.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* diagnosis of Crohn's Disease (CD) or Ulcerative Colitis (UC) with mild to moderate colitis for at least 6 months (CD: Harvey-Bradshaw-Index Score 5-16; UC: Partial Mayo Score 2-6)
* stable IBD-specific medication dosage for at least 3 months [such as 5-aminosalicylates (5-ASA), thiopurines or biologicals (therapeutic antibodies such as infliximab, adalimumab, vedolizumab, etc.)]
* inpatient admission to the Department for Internal and Integrative Medicine at the Sozialstiftung Bamberg, Germany for regular treatment
* clinical indication and performance of an initial colonoscopy with confocal laser endomicroscopy (CLE)
* signed informed consent form

Exclusion Criteria:

* IBD without inflammation of the colon (e.g. Crohn's Disease without colitis)
* active flare of IBD
* CRP ≥ 100 mg/l
* artificial bowel outlet in front of the colon (ileostomy)
* high regular consumption of blueberries (≥ 300 g cultivated blueberries or ≥ 150 g wild blueberries per week) or administration of blueberry therapy in the last 3 months
* participation in another therapeutic study within the last 30 days
* Known intolerance to blueberries or their ingredients such as contained anthocyanins or fructose (e.g. fructose malabsorption)
* presence of known serious infectious diseases e.g. of the liver such as HIV, hepatitis B and C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of the intestinal inflammation status evaluated via fecal calprotectin levels | week 0, 12, 24
  The inflammation status is evaluated through measurement of fecal calprotectin levels in stool samples. This biomarker provides information about the inflammatory status in the intestine and serves as an objective measure of disease activity.

SECONDARY OUTCOMES:
Improvement of Crohn's disease severity evaluated by Harvey-Bradshaw-Index (HBI) | week 0, 12, 24
  The disease severity of CD patients is evaluated via a validated questionnaire that is specific for Crohn's Disease (Harvey-Bradshaw-Index):
  The HBI was designed as a simplified version of the CDAI to enable systematic collection of clinical data on Crohn's disease and is used to assess the degree of illness in individuals with Crohn's disease. The index considers five, exclusively clinical parameters. A specific score is assigned for each parameter. To assess disease activity, the sum score is formed from questions on general condition, abdominal pain, number of unformed bowel movements per day, abdominal resistance and complications. The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
Improvement of ulcerative colitis disease severity evaluated by MAYO-Score | week 0, 12, 24
  The disease severity of UC patients is evaluated via a validated questionnaire that is specific for ulcerative colitis (MAYO-Score): The Mayo Score is the most commonly used scoring system for UC in clinical trials and routine practice. It was developed to standardize the severity of a patient's UC symptoms, which is particularly helpful to assess response to treatment over time. For this study, the partial MAYO-Score is applied, which comprises only the non-invasive components of the full Mayo score. Endoscopic findings are not taken into account. The index considers three clinical parameters, each of which is assigned a score from 0 to 3 leading to a maximum score of 9 points. Clinical response is defined as a decrease of at least 2 points.
Evaluation of IBD-SI (Inflammatory Bowel Disease Symptom Inventory) | week 0, 12, 24
  The IBD-SI combines items from existing clinician-rated or diary-format inventories. After factor analysis, 38 items were retained on 5 subscales: bowel symptoms, abdominal discomfort, fatigue, bowel complications, and systemic complications. A total score as well as subscale scores will be calculated.
Evaluation of disease-specific quality of life by IBD-Q (Inflammatory Bowel Disease Questionnaire) | week 0, 12, 24
  The IBD-Q is the most frequently used questionnaire for disease-specific quality of life in clinical studies on Crohn's disease. It operationalizes quality of life on 4 dimensions (emotional and social impairment as well as bowel-related and systemic symptoms), in addition to a sum score. Answers are recorded on a 7-point Likert scale. High values mean good, low values a reduced quality of life (1=worst score, 7=best score). The total IBD-Q scale ranges from 32 to 224. A score of ≥ 170 can be considered as normal quality of life.
Assessment of health-related quality of life with the Short Form 12 Health Survey (SF-12) | week 0, 12, 24
  The Short Form 12 Health Survey (SF-12) is a validated tool with 12 questions for the general assessment of the physical and mental health status of patients that is widely used in clinical studies. It is the shorter version of the SF-36 questionnaire. Two scores - one score for the physical component (PCS) and one score for the mental component (MCS) - represent the results. The SF-12 physical scale score represents general health perception, physical functioning, physical role functioning, and pain. The mental health score reflects emotional role functioning, mental well-being, negative affectivity, and social functioning. The questionnaire has already been used in various medical publications in different disciplines due to its wide range of applications. A low total value correlates with a poor quality of life, a higher one with a better one. The values determined are compared with the values of the normal population.
Assessment of the severity of the fatigue syndrome with the Multidimensional Fatigue Inventory (MFI-20) | week 0, 12, 24
  The Multidimensional Fatigue Inventory (MFI) is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity and mental fatigue. The German validated version is used. A scale from 1 to 7 is used to indicate how aptly certain statements regarding fatigue represent the participants' experiences. Higher total scores correspond with more acute levels of fatigue.
Assessment of perceived stress using the Perceived Stress Scale (PSS-10) | week 0, 12, 24
  The Perceived Stress Scale (PSS-10) is a well-established self-report scale and an international standard instrument for measuring perceived stress. The ten questions ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way on a five-point scale from 'never' to 'very often'. The PSS score is obtained by summing across all items after responses to the four positively stated items have been reversed. Higher scores indicate higher levels of perceived stress.
Assessment of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS) | week 0, 12, 24
  Anxiety and depression are measured using the Hospital Anxiety and Depression Scale (HADS). The HADS was developed specifically for physically ill patients in clinical settings. The questionnaire contains 14 items: 7 on the anxiety and 7 on the depression scales. The sum values of the HADS-A (anxiety) and HADS-D (depression) scales lie in the 0-21 range, with higher values indicating a stronger manifestation of anxiety/depressiveness. The German validated version is used.
Assessment of food-related quality of life using the FR-QoL-29 questionnaire | week 0, 12, 24
  A validated questionnaire for the systematic assessment of food-related quality of life (FR-QoL) in IBD patients is used to assess psychosocial factors in connection with eating and drinking, such as enjoying food, managing restrictions, and maintaining social relationships. The FR-QoL-29, which contains 29 items, each scored on a 5-point Likert scale (1 = strongly agree; 2 = agree; 3 = neither agree nor disagree; 4 = disagree; 5 = strongly disagree), with 4 questions reversed for scoring. Scores are summed, with a total possible score ranging from 29 to 145, where higher scores reflect a greater FR-QoL.
Assessment of frequency of consumption and usual portion sizes of particular food groups using the DEGS-Food Frequency Questionnaire | week 0, 4, 8, 12, 16, 20, 24
  A food frequency questionnaire (FFQ) is used to determine the frequency of consumption and usual portion sizes of a total of 53 food groups consumed in the last four weeks. The dietary questionnaire was developed and validated for the use in the German Health Examination Survey for Adults 2008-2011 (DEGS). In this study it is used to assess whether the participants' dietary habits change throughout the study and whether they apply the diet taught during nutritional therapy at the inpatient stay at the clinic for internal and integrative medicine in Bamberg.
Patient Diary | week 0 to week 24
  Over the course of the study, the participants keep a diary in which they document their daily blueberry intake and symptoms to enable the evaluation of their compliance and their tolerance of the blueberry powder.
Colonoscopy/Sigmoidoscopy with confocal laser endomicroscopy (CLE) | week 0, 12, 24
  At week 0, participants undergo a colonoscopy with confocal laser endomicroscopy (CLE) when clinically indicated as part of their inpatient care. Thereby, the inflammatory status and the intestinal barrier is routinely analyzed. Participants return for a voluntary colonoscopy or sigmoidoscopy at week 12 and week 24. Confocal laser endomicroscopy (CLE, Cellvizio System from Mauna Kea Technology) is the first technology that enables live characterization of the intestinal mucosa and barrier integrity at the cellular level during endoscopy at up to 1000x magnification, allowing local intestinal barrier disorders to be identified and targeted biopsies to be taken. This combined examination of endoscopy and CLE thus enables a comprehensive assessment of the intestinal mucosa on a macroscopic, microscopic and functional level in real time.
Histopathological analysis of ileo-colorectal biopsies | week 0, 12, 24
  Intestinal biopsies, which are routinely taken during colonoscopy/sigmoidoscopy, are processed for histopathological analysis of the mucosal and epithelial structure as well as of the immune cell compartment (H&E staining).
Immunohistochemical analysis of ileo-colorectal biopsies | week 0, 12, 24
  Intestinal biopsies, which are routinely taken during ileocolonoscopy, are stained using immunohistochemistry and examined for the expression of specific marker proteins. For example, the intestinal barrier will be examined by immunohistochemical analysis of the tight junction marker proteins occludin and claudin-2 or the migration of specific immune cells such as T-lymphocytes using CD3 staining.
Gene expression analysis of ileo-colorectal biopsies | week 0, 12, 24
  Intestinal biopsies taken in addition to those routinely taken during ileocolonoscopy are used for transcriptional analysis by q-PCR to study the gene expression of particular immune cell or inflammatory marker proteins as well as tight junction proteins.
Evaluation of the systemic inflammatory status by analysis of serum-cytokine concentrations | week 0, 12, 24
  To evaluate the systemic inflammatory status, the level of various cytokines such as IL-1β, IL-6, IL-8, IL-10, TNF, IFN-γ, IL-17or IL-4 is analyzed in the serum.
Complete blood count | week 0, 12, 24
  A complete blood count including iron status and liver markers is made. It provides information about the number and type of immune cells. In combination with the general inflammatory markers C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR), the complete blood count allows conclusions about the presence and extent of systemic inflammation as well as the disease activity. Checking the iron status and liver markers can provide indications of IBD-associated complications such as anemia and liver dysfunction.
C-reactive protein (CRP) in the blood | week 0, 12, 24
  The concentration of the inflammation marker CRP is measured in the blood.
Erythrocyte Sedimentation Rate (ESR) | week 0, 12, 24
  Determination of the ESR of the blood.
Analysis of inflammatory markers in the stool | week 0, 12, 24
  Besides Calprotectin, also the concentrations of other inflammatory markers such as Lactoferrin and PMN-Elastase are analyzed in the stool to evaluate the intestinal inflammation status quantitatively.
Analysis of fecal biomarkers to evaluate the integrity of the intestinal barrier | week 0, 12, 24
  The concentrations of fecal biomarkers such as Zonulin or α-1-Antitrypsin are determined to quantitatively evaluate the integrity of the intestinal barrier.
Determination of the I-FABP concentration in the serum | week 0, 12, 24
  The I-FABP concentration is measured in serum samples to evaluate the intestinal permeability. I-FABP is a protein exclusively found in intestinal epithelial cells. If the intestinal epithelium is damaged, I-FABP is released into the circulation and can be measured in the serum. Therefore, I-FABP serum levels are a valid biomarker for intestinal permeability in coeliac disease, wheat sensitivity and also in inflammatory bowel disease.
Determination of the fecal β-Defensin concentration | week 0, 12, 24
  Fecal concentrations of the antimicrobial peptide β-Defensin are determined in the stool.
Fecal microbiome analysis | week 0, 12, 24
  The fecal microbiome is analyzed in stool samples in order to determine the influence and the prebiotic properties of the blueberry-rich diet on the intestinal microbiome.
Analysis of fecal metabolites | week 0, 12 and 24
  Microbial metabolites such as short chain fatty acids (SCFAs) are analyzed in stool samples in order to determine the influence and the prebiotic properties of the blueberry-rich diet on the intestinal microbiome. Prebiotics are nutritional components that promote the growth and activity of beneficial bacterial species. Prebiotics serve as a nutritional basis for these bacteria and promote, for example, their production of SCFAs that act as essential energy substrates for enterocytes and immune cells. These metabolites have been shown to influence immune cell maturation, immune homeostasis, host energy metabolism and the maintenance of mucosal integrity. Therefore, the combined evaluation of microbiome and microbial metabolites in the stool can contribute to a better understanding of the interplay of these factors in the development and treatment of IBD.
Metabolite profiling in the urine | week 0, 12 and 24
  Metabolite profiling is done from urine samples. This can also provide valuable insights into the (dys)regulation of gut microbial metabolism and host-microbe co-metabolism in the context of IBD.
Analysis of oxidative stress in the urine | week 0, 12, 24
  8-hydroxy-2-deoxyguanosine (8-OHdG) is analyzed in urine samples as a marker for oxidative stress in order to evaluate the antioxidant potential of the blueberry-rich diet. Oxidative stress plays an important role in a variety of chronic inflammatory diseases, including IBD. Oxidative stress describes a disturbance in the balance between the production and accumulation of reactive oxygen species (ROS). ROS are scavenged by the antioxidant system but can oxidize proteins, lipids and DNA in excessive concentrations. Resulting DNA damage is normally repaired and the oxidation products are excreted in the urine. 8-OHdG, a product of DNA guanine residue oxidation by ROS is an established biomarker for oxidative damage to DNA. Blueberries are known for their antioxidant potential. To evaluate the influence of a blueberry-rich diet on oxidative stress and antioxidant potential, 8-OHdG is analyzed in urine samples.
Analysis of the antioxidant capacity in the serum | week 0, 12, 24
  In addition to the evaluation of oxidative stress in the urine, the systemic antioxidant capacity of the blood is analyzed in serum samples as a reduced total antioxidant capacity can reflect the clinical disease activity.
Analysis of the thiol status in the serum | week 0, 12, 24
  The thiol status records the protective, free thiol groups that intercept extracellular radicals and bind toxic metals and pollutants. The thiol status is therefore a parameter of the extracellular protective system. Reduced thiol levels promote oxidative stress and serve as a marker for chronic inflammatory processes.
Analysis of the peroxidation of lipids in the serum | week 0, 12, 24
  The peroxidation of lipids is evaluated in the serum. The determination of lipid peroxides can indicate an imbalance in antioxidant homeostasis.
  Lipid peroxides are formed by the reaction of free radicals (ROS) with lipid structures, whereby unsaturated fatty acids contained in lipid membranes or lipid vesicles are oxidized. An excess of lipid peroxides is associated with chronic inflammatory processes.
Analysis of the composition of bile fluid | week 0, 12, 24
  In case an esophagogastroduodenoscopy is performed as part of the routine inpatient care, a sample of bile fluid is collected by simple aspiration from the duodenum in order to assess the secretion and composition of bile acids and their metabolites. Bile acids and their metabolites can have a significant impact on gut health in IBD patients. They have the capacity to modulate inflammation, alter the microbiome and affect the intestinal barrier integrity by regulating the expression of tight junction proteins that control the permeability of the gut wall.
Anamnesis | week 0, 12, 24
  Data collected during anamnesis in the course of the routine in-patient stay such as the course of disease or working ability are documented to enable an evaluation of the participants' medical condition and health status.
Concomitant medication | week 0, 12, 24
  Concomitant medication and especially CED-related therapy of the study participants is documented throughout the study.
Medical history | week 0, 12, 24
  Information on concomitant diseases and the medical history of the study participants is routinely collected and recorded in the course of the in-patient stay as well as in the course of the study to evaluate the participants' medical condition and health status.
Social demographics | week 0
  Social demographic aspects are collected in order to describe the patient collective of the study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Univ. Prof. Dr. med., Principal Investigator — Universität Duisburg-Essen
Locations (1):
- Sozialstiftung Bamberg, Bamberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No